CLINICAL TRIAL: NCT01418300
Title: Comparison of Conventional Triple Therapy Versus Sequential Therapy for H. Pylori in Peptic Ulcer Disease: Prospective Randomized Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jun-Won Chung (Industry)
Responsible Party: Sponsor-Investigator, Jun-Won Chung, principal investigator, Jeil Pharmacy Co.
Organization: Jeil Pharmacy Co. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMC2010-088
Record Dates: First submitted 2011-08-13; First posted 2011-08-17 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2011-08

CONDITIONS: Helicobacter Infected Patients

ARMS (2):
- sequential therapy (Active Comparator): first five day amoxicillin+PPI later five day PPI+clarithromycin+metronidazole
  Interventions: Drug: sequential versus triple
- conventional triple thearpy (Active Comparator): PPI+amoxicillin+clarithromycin
  Interventions: Drug: sequential versus triple

INTERVENTIONS:
Drug: sequential versus triple — sequential: lansoprazole 30mg bid+amoxicillin 100mg bid for first five day lansoprazole 30mg bid+clarithromycin 500mg bid+metronidazole 500mg for 5day conventional tripe lansoprazole 30mg bid+clarithromycin 500mg bid+amoxicillin 1000mg bid

SUMMARY:
The purpose of this study is to improve first line Helicobacter pylori eradication rate and to compare the sequential versus conventional triple therapy.

ELIGIBILITY:
Inclusion Criteria:

* peptic ulcer diseae
* two test positive rapid urease test, culture, histology

Exclusion Criteria:

* lactating or pregnant
* previous stomach surgery
* severe underlying disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
the eradication rate by urea breath test | 4-6 week later after completion of therapy
  to compare the eradication rate (intention-to-treat and per protocol) by urea breath test at least four weeks after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Gil Medical Center, Incheon, South Korea